CLINICAL TRIAL: NCT01901042
Title: Efficacy of Symbiotic in the Reduction of Acute Radiation Proctitis Symptoms. A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Efficacy of Symbiotic in the Reduction of Acute Radiation Proctitis Symptoms
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Federal University of Mato Grosso (Other)
Responsible Party: Principal Investigator, Jose Eduardo de Aguilar-Nascimento, MD, PhD, Federal University of Mato Grosso
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: marianan
Record Dates: First submitted 2013-05-26; First posted 2013-07-17 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: Radiation Proctitis; Prostate Cancer
Keywords: Quality of life; Symbiotic; Proctitis/Radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms; Proctitis | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Symbiotic (Experimental): Patients in this group received sachets with a symbiotic product in powder form containing 4.3 g of dietary fiber and Lactobacillus reuteri in a concentration greater than 1.0 x 108 colony forming units (CFU), with five grams per sachet (Fibermais Flora Nestlé Brazil).
  Interventions: Dietary Supplement: Symbiotic
- Maltodextrin (Placebo Comparator): patients in this group received sachets five grams of maltodextrin per sachet with identical casing and identical aspect to the product of the other arm group, and were instructed to proceed in the same way as those of the symbiotic group
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Symbiotic — Sachets with a symbiotic product in powder form containing 4.3 g of dietary fiber and Lactobacillus reuteri in a concentration greater than 1.0 x 108 colony forming units (CFU), with five grams per sachet (Fibermais Flora Nestlé Brazil).
  Other Names: FiberMais Flora (Nestlé, Brazil)
  Arms: Symbiotic
Dietary Supplement: Maltodextrin — Control patients will receive sachets containing maltodextrin
  Other Names: Placebo supplement
  Arms: Maltodextrin

SUMMARY:
Radiation proctitis is quite common in treatment of pelvic tumors. We investigated whether the use of symbiotic would prevent early symptoms of radiation proctitis and improve the quality of life in patients undergoing radiotherapy for prostate cancer treatment. We randomized patients to intake one sachet of either a symbiotic product containing 4.3 g of dietary fiber and Lactobacillus reuteri in a concentration greater than 10(8)colony forming units (CFU)(Fibermais Flora Nestlé Brazil) or sachets containing 5 g of maltodextrin. They were instructed to dilute one sachet in 200mL of water and drink once a day during the week before the beginning of radiotherapy sessions, and increase the dose to two sachets daily after the beginning of the sessions for four weeks. Every week a questionnaire named EORTC QLQ-PRT23 was applied to evaluate GI symptoms and quality of life.

DETAILED DESCRIPTION:
This is a prospective randomized, double-blind, placebo-controlled trial. The study included consecutively 20 patients referred for treatment of prostate cancer using three-dimensional conformal radiotherapy (3D-RCT). All patients who agreed to participate signed an informed consent form. The exclusion criteria used in this study were: a patient's refusal to participate in the research and history of surgery involving the rectum or inflammatory bowel disease Patients were randomly assigned to receive sachets containing either a symbiotic product in powder form containing 4.3 g of dietary fiber and Lactobacillus reuteri in a concentration greater than 1.0 x 108 colony forming units (CFU), with five grams per sachet (Fibermais Flora Nestlé Brazil) (symbiotic group) or maltodextrin (5g) with identical casing and identical aspect of the symbiotic group. All subjects were instructed to dilute one sachet in a glass of water and drink once a day during the week before the beginning of radiotherapy sessions, increasing the dose to two sachets daily after the beginning of the sessions.

EORTC QLQ-PRT23 questionnaire Each participant answered the questions of the EORTC QLQ-PRT23 questionnaire before the beginning of radiotherapy and immediately after the first, second, third and fourth weeks of treatment. The questions were always asked by an examiner blinded to the study design and type of treatment used. The EORTC QLQ-PRT23 questionnaire, originally developed in English, was translated into Portuguese following the protocol described at the EORTC Translation Procedure : The sum of points obtained by each patient through the first 21 questions of the EORTC QLQ-PRT23 was recorded. All these 21 questions received a number of points according to the intensity of each symptom or problem during the previous week, as follows: - "Not at all" = 1 point; "A little" = 2 points; "Quite a bit" = 3 points; and "Very much" = 4 points.

Radiotherapy protocol A total dose of 66-76 Gy during 6-8 weeks was programmed for each individual. Patients were followed-up until the fourth week of radiotherapy and the cumulative dose of radiation was compared weekly between the two groups. Each patient was scheduled to receive a dose of two grays (Gy) per day, from Monday to Friday with weekend interval, totaling 10 Gy per week and 40 Gy after the 4th week of treatment. The irradiated rectal volume after an accumulated dose of 40 Gy was compared between the two groups using dose-volume histograms and presented in percentages of the rectal volume which received 10 Gy (V10), 20 Gy (V20), 30 Gy (V30), and 40 Gy (V40).

Outcome variables The endpoints of the study were the intensity of the gastrointestinal symptoms and quality of life. All patients were scored with the sum of questions from 1 to 21 to represent both gastrointestinal symptoms and quality of life; and the sum of the scores obtained with questions numbered from 1 to 15, which refer only to gastrointestinal symptoms. Presence of blood in stools and tenesmus intensity were also assessed according to the score described above and used in the questionnaire. It was also recorded the maximum number of evacuations that each patient had over a period of 24 hours each week.

Statistical analysis For the calculation of the sample, it was estimated that the symbiotic group would present a median of four points lower than the score of the placebo group over four weeks. A total of twenty patients (10 in each group) was calculated considering an error alpha of 1% and a beta error of 90%. The Statistical Package for Social Sciences (SPSS) for Windows 9.0 was used for statistical analysis. A level of 5% (p <0,05) was established for significance. Fischer's test or chi-square test was used for categorical variables. For continuous data, we used the Mann-Whitney or Student's t according to the homogeneity (Levene test) and normality (Kolgomorov-Smirnov test) data. Repeated measures ANOVA was used to analyze the responses obtained by the EORTC QLQ-PRT23 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing radiotherapy due to prostate cancer

Exclusion Criteria:

* refuse to participate, previous rectal condition or surgery, inflammatory bowel disease

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Changes in gastrointestinal symptoms | once a week during five weeks
  Patients responded to a questionnaire (EORTC QLQ-PRT23)on their gastrointestinal symptoms every week during five weeks. One week before and four weeks during their radiotherapy program we looked at the changing in gastrointestinal symptoms
Changes in quality of life | once a week during five weeks
  Patients responded to a questionnaire (EORTC QLQ-PRT23)on their quality of life every week during five weeks. One week before and four weeks during their radiotherapy program we looked at changing in quality of life

CONTACTS AND LOCATIONS:
Overall Officials: JOSE E AGUILAR-NASCIMENTO, MD, PhD, Principal Investigator — Federal University of Mato Grosso